CLINICAL TRIAL: NCT00252915
Title: Reconstruction of Monocytic Immunocompetence by Granulocyte-macrophage-colony Stimulating Factor (GM-CSF) in Patients With Severe Sepsis and Septic Shock: a Prospective, Randomised, Double-blind, Placebo-controlled Study
Brief Title: Reconstruction of Monocytic Immunocompetence by Granulocyte-macrophage-colony Stimulating Factor (GM-CSF) in Patients With Severe Sepsis and Septic Shock
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Charite University Medicine Berlin, Charite
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GM-CSF-1
Record Dates: First submitted 2005-11-14; First posted 2005-11-15 (Estimated); Last update posted 2011-05-26 (Estimated); Status verified 2009-07

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Verum (Experimental): GM-CSF therapy
  Interventions: Biological: GM-CSF (verum)

INTERVENTIONS:
Biological: GM-CSF (verum) — sagramostim

SUMMARY:
There is basic science evidence that GM-CSF reconstructs cellular immunity in septic patients. In this prospective, randomised double-blind, placebo-controlled trial, we investigate whether this can be achieved in patients with severe sepsis and septic shock.

DETAILED DESCRIPTION:
GM-CSF reconstructs cellular immunity in septic patients. In this prospective, randomised double-blind, placebo-controlled trial, we investigate whether this can be achieved in patinets with severe sepsis and septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Severe sepsis or septic shock,
* Presence of infection,
* 2 SIRS criteria,
* Acute organ dysfunction,
* Immunoparalysis,
* Informed consent

Exclusion Criteria:

* Pregnancy,
* Known allergies to study medication or components,
* Moribound patient,
* Autoimmune disease,
* HIV-infection,
* Acute MI or pulmonary embolism,
* Cpr during last 72 hours,
* Patients who participate in a different clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2005-11; Primary Completion 2007-01 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
reconstitution of monocytic immunity as defined as a mHLA-DR expression >15,000 molecules per cell at study day 9 | after therapy

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Dieter Volk, MD, Study Chair — Charite University, Berlin, Germany; Joerg C Schefold, MD, Principal Investigator — Charite University Medicine; Christian Meisel, MD, Principal Investigator — Charite University Medicine

REFERENCES:
- [Derived] Meisel C, Schefold JC, Pschowski R, Baumann T, Hetzger K, Gregor J, Weber-Carstens S, Hasper D, Keh D, Zuckermann H, Reinke P, Volk HD. Granulocyte-macrophage colony-stimulating factor to reverse sepsis-associated immunosuppression: a double-blind, randomized, placebo-controlled multicenter trial. Am J Respir Crit Care Med. 2009 Oct 1;180(7):640-8. doi: 10.1164/rccm.200903-0363OC. Epub 2009 Jul 9. PMID 19590022